CLINICAL TRIAL: NCT03442270
Title: Detection Rate of Serrated Adenomas in the Screening Colonoscopy Population
Brief Title: Detection Rate of Serrated Adenomas in Screening Colonoscopy
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Collaborators: TriHealth Hatton Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17-074
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-05

CONDITIONS: Healthy Patients Undergoing Screening Colonoscopy
Keywords: Serrated Adenoma, Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — This is an observational study, so standard of care will be followed.

SUMMARY:
An observational prospective will be conducted to determine the detection rate of serrated adenoma during screening colonoscopy at our institution. Additionally, the variability of serrated adenoma detection among endoscopists will be evaluated and the characteristics of serrated adenomas will be described.

DETAILED DESCRIPTION:
Colonoscopy screening is a preventative measure for colorectal carcinoma (CRC), a highly malignant and dangerous cancer. Extensive research on the adenoma detection rate has provided national standards and quality metrics to help assess competence of endoscopists. Currently, there are no standards established for serrated adenomas. The proposed study would be conducted at Good Samaritan Hospital (GSH) and TriHealth Surgery Center West. This is an observational study and does not involve any patient interventions. However, because patient healthcare data will be collected for research, informed consent will be obtained shortly before the procedure. The main study objective is to determine the detection rate of serrated adenoma during screening colonoscopy at our institution. Additionally, the variability of serrated adenoma detection among endoscopists will be evaluated and the characteristics of serrated adenomas will be described.

ELIGIBILITY:
Inclusion Criteria:

* Males and females

Exclusion Criteria:

* First degree relative (patient's parent, sibling or child) diagnosed with colorectal carcinoma at age of 59 or under
* New onset of iron deficiency anemia (within past 3 months)
* Abnormal imaging of colon within past 3 months
* Inadequate visualization reported by endoscopist
* Pregnant women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients 50 years or older undergoing first-time colonoscopy screening
Sampling Method: Non-Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Serrated Adenoma | March 2018 to October 2018
  Prevalence of Serrated Adenoma

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim HY, Kim SM, Seo JH, Park EH, Kim N, Lee DH. Age-specific prevalence of serrated lesions and their subtypes by screening colonoscopy: a retrospective study. BMC Gastroenterol. 2014 Apr 28;14:82. doi: 10.1186/1471-230X-14-82. PMID 24775268